CLINICAL TRIAL: NCT02604394
Title: Rheolytic Thrombectomy in Patients With Acute STEMI and Large Thrombus Burden
Acronym: Rheo-STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Magdi Yacoub Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rheo-STEMI
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: ST Elevation Myocardial Infarction; STEMI
Keywords: Rheolytic Thrombectomy; Percutaneous Coronary Intervention; Angioplasty; Cardiac Magnetic Resonance Imaging; Myocardial Salvage Index; STEMI, ST elevation Myocardial Infarction; Corrected TIMI Frame Count, cTFC; Index of microcirculatory resistance, thermodilution, IMR
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rheolytic Thrombectomy with PCI (Active Comparator): Rheolytic Thrombectomy (RT) will be performed with the The AngioJet rheolytic thrombectomy system (Medrad Interventional/Possis, Minneapolis, Minnesota).
  The single-pass antrograde thrombectomy technique will be used.
  Interventions: Procedure: Rheolytic Thrombectomy; Procedure: Conventional PCI
- Conventional PCI (Sham Comparator): In patients in the conventional PCI group, antegrade flow in the culprit vessel will be established with conventional PCI with preference of direct stenting and use of manual thrombus aspiration when deemed necessary by the operator.
  Interventions: Procedure: Conventional PCI

INTERVENTIONS:
Procedure: Rheolytic Thrombectomy — RT will be performed with the The AngioJet rheolytic thrombectomy system (Medrad Interventional/Possis, Minneapolis, Minnesota).
  The RT system includes three units: disposable catheter, disposable pump set and a reusable drive unit:
  1. The single-use catheter has two lumens; one allows for the in-flow of high velocity saline jets through the catheter tip, and the other allows for the evacuation of thrombotic debris and passage of a guidewire.
  2. The disposable pump connects to a bag of heparinized saline.
  3. The drive unit pumps pressurized heparinized saline at 10,000 psi at the tip of the catheter,
  Other Names: The AngioJet rheolytic thrombectomy system; AngioJet
  Arms: Rheolytic Thrombectomy with PCI
Procedure: Conventional PCI — In patients in the conventional PCI group, antegrade flow in the culprit vessel will be established with conventional PCI with preference of direct stenting and use of manual thrombus aspiration when deemed necessary by the operator.
  Other Names: Percutaneous Coronary Intervention

SUMMARY:
Coronary obstruction by an occlusive thrombus complicating a ruptured or eroded atherosclerotic plaque is the most frequent pathologic substrate of acute myocardial infarction (AMI).

Timely restoration of perfusion and thereby myocardial salvage is the single most important objective in the management of patients with ST segment-elevation myocardial infarction (STEMI).

To address these uncertainties, our study aims to evaluate the role of RT in patients who are most likely to benefit from it (thrombus grade 4 and 5) using a sensitive, quantitative, and reproducible parameter; CMR-derived myocardial salvage. also, to determine whether Rheolytic Thrombectomy (RT) before conventional PCI to the culprit vessel as compared to conventional PCI (with or without MTA) results in improved myocardial salvage; and to identify clinical and angiographic determinants of any difference observed between both treatment groups.

DETAILED DESCRIPTION:
Coronary obstruction by an occlusive thrombus complicating a ruptured or eroded atherosclerotic plaque is the most frequent pathologic substrate of acute myocardial infarction (AMI) , , . Timely restoration of perfusion and thereby myocardial salvage is the single most important objective in the management of patients with ST segment-elevation myocardial infarction (STEMI).

Primary percutaneous coronary intervention (PCI) is now the preferred treatment for STEMI patients and is effective in opening the infarct-related artery (IRA) and restoring Thrombolysis in Myocardial Infarction (TIMI) III flow in more than 95% of patients , , . However the presence of a large thrombus burden increase the incidence of adverse outcomes including persistent or transient no-reflow and in-hospital major adverse cardiac events (MACEs), possibly due to distal atherothrombotic embolization, with ensuing disruption of the microvascular network and failure of myocardial reperfusion . The microvascular obstruction occurs in 10% of STEMI patients with a patent epicardial vessel after primary PCI , , . It is associated with an increased infarct size, reduced recovery of ventricular function, and increased mortality , , , , , , .

Removal of thrombi from the IRA during primary PCI may prevent distal embolization and improve myocardial perfusion and thus long term clinical outcomes. However studies conducted to date provide mixed results , , , , , .The two largest randomized trials to date comparing manual thrombus aspiration (MTA) followed by PCI to PCI only are the Thrombus Aspiration during PCI in Acute Myocardial Infarction (TASTE) study , and Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction (TAPAS) study , . They further illustrate the existing uncertainties.

TAPAS study showed improvement of the myocardial blush grade (primary endpoint) and reduction of cardiac mortality at one year follow up in patients of the MTA group compared to those in the conventional-PCI group. However, it is important to note that TAPAS was not powered to detect differences in clinical outcome. TASTE study showed no mortality benefit of MTA at one year follow up. These results concluded that routine use of thrombus aspiration is not supported by current evidence however, selective use may improve tissue perfusion in some patients .Accordingly MTA is currently a class IIb recommendation in the European Society of Cardiology (ESC) guidelines for myocardial revascularization in STEMI patients , and a class IIa recommendation in the 2013 ACC/AHA STEMI guidelines . The latter was released before the results of TASTE were published.

MTA is ineffective in ≈30% of patients. Furthermore, residual thrombi after MTA are present in virtually all patients when studied by optical coherence tomography (OCT).27, . The currently existing alternative technique for removal of intracoronary thrombi is the Rheolytic Thrombectomy (RT) by Angiojet device. RT is a catheter-based system that utilizes multiple high-velocity, high-pressure saline jets introduced through orifices in the distal tip of the catheter to create a localized low-pressure zone (Venturi-Bernoulli effect), resulting in a vacuum effect with the entrainment and dissociation of bulky thrombi. The jets break down thrombi into small particles and propel them proximally through the exhaust lumen, leading to the aspiration and removal of thrombotic debris without embolization.

The two largest randomized trials to date studying the benefits of RT in patients presenting with acute STEMI are (JETSTENT) Study and (AIMI) study.

In the JETSTENT study8, ST-segment resolution was more frequently achieved in the RT arm. There were fewer MACEs (death, MI, target vessel revascularization, and stroke) in the RT arm at 12 months (p=0.036). Infarct size at one month did not differ between both arms. However, results of JETSTENT need to be interpreted with caution; in the strict statistical sense, it was a negative trial. Studies with a co-primary endpoint require a p value of 0.05 for both endpoints or 0.025 for a single endpoint. This was not achieved in JETSTENT. However, multivariable analysis showed that the use of rheolytic thrombectomy was independently associated with improved clinical outcomes at one year - acknowledging that that latter was not one of the primary endpoints.

On the other hand, in the AIMI 24 , the final infarct size was higher in the adjunct RT group compared to PCI only group. Final TIMI III flow was lower in the adjunct RT group. Thirty-day MACEs were higher in the adjunct RT group, a difference primarily driven by very low mortality rates in patients treated with PCI only. There were no significant differences in TIMI blush grade or ST-segment resolution between both groups. However, there are several limitations to AIMI; a) the study did not require angiographic evidence of thrombus, and in fact, excluded patients with very large thrombus burden, b) a retrograde technique - which involves crossing the lesion before activation of the device - was used in the majority of patients in the RT group, c) the time delay between admission and use of RT (door-to-device) was very long, d) compared to the RT group, more patients in the PCI-only group had baseline TIMI III flow (44% vs. 63%, p= 0.05). Collectively, these factors might have overshadowed any potential benefit of RT in AIMI.

In another study, Parodi et al 31, compared MTA to RT in patients with acute STEMI using residual thrombus burden (assessed by OCT) as the primary endpoint. The study did not meet the primary end point; the number of OCT quadrants containing residual thrombus .However, angiographic thrombus grade decreased significantly after RT, and all markers of reperfusion (secondary endpoints) were better in the RT arm. There was a trend toward higher rate of early ST-segment elevation resolution in the RT arm as compared with the MTA arm. These findings suggest that RT may be more effective than MTA but to a lesser degree than hypothesized by the investigators. Furthermore, calculation of thrombus volume by OCT is extremely challenging given the inability to accurately define the border between disrupted atherosclerotic plaques and superimposed thrombi, which is further blurred by the optical shadowing of red thrombus.

To address these uncertainties, our study aims to evaluate the role of RT in patients who are most likely to benefit from it (thrombus grade 4 and 5) using a sensitive, quantitative, and reproducible parameter; CMR-derived myocardial salvage. CMR Cardiac MRI can provide a wide range of information such as myocardial edema (myocardium at risk), microvascular obstruction (MVO), location and "transmurality" of necrosis, as well as quantification of infarct size . Moreover, CMR provides accurate and reproducible measurements of ventricular volumes and function. For these reasons, cardiac MRI is currently perceived as the ideal tool for evaluation of global post-infarction remodeling.

Myocardial edema in the acute phase of myocardial infarction can be visualized as a bright signal on T2-weighted images, defining 'myocardium at risk .The major advantages of this technique are distinguishing chronic from acute infarction, and quantifying the proportion of myocardial salvage assessed retrospectively by comparing T2-weighted edematous (at risk) size and late gadolimium enhancement (LGE) images (scar). LGE images are T1-weighted inversion recovery sequences acquired about 10 min after intravenous administration of gadolinium and the inversion time is chosen to null myocardial signal using 'inversion time scout' or 'look locker' sequences .

Delayed post-contrast sequences are currently used also to evaluate persistent microvascular dysfunction/damage: in the context of white LGE regions (infarcted myocardium) dark hypoenhanced areas may coexist, traditionally referred to as microvascular obstruction. Microvascular obstruction has been initially defined as hypo enhancement at 1-2 min after gadolinium injection; the final infarct size depends mainly on the extent of the so-called 'risk area', defined as the myocardial area related to an occluded coronary artery with complete absence of blood flow, either antegrade or collateral .

These novel CMR-derived parameters have emerged as potential indices of adverse remodeling, with the most attractive being myocardial salvage. Myocardial salvage is a prognostically validated therapeutic target in primary PCI , , , , with myocardial salvage index being a strong predictor of major cardiac events and mortality at 6-month . Myocardial salvage is defined as the difference between the initial jeopardized area at risk (determined by T2-weighted MRI) at baseline and final infarct size (determined by contrast-enhanced MRI). The myocardial salvage index is defined as final infarct size indexed to the initial area at risk , , .

Objectives of the study:

1. To determine whether Rheolytic Thrombectomy (RT) before conventional PCI to the culprit vessel as compared to conventional PCI (with or without MTA) results in improved myocardial salvage.
2. To identify clinical and angiographic determinants of any difference observed between both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* STEMI with time from symptom onset of <12 hours duration.
* STEMI with time from symptom onset < 24 hours, in the presence of ongoing ischaemia, life-threatening arrhythmias or if pain and ECG changes have been stuttering.

Exclusion Criteria:

* Clinical exclusion criteria:

  1. STEMI patients receiving fibrinolytic therapy.
  2. Cardiogenic shock.
  3. Patients with clinical, hemodynamic, or electrical instability as well as those judged to be critically ill or when there is need to minimize the procedure length to the shortest possible time.
  4. Patients refusing to participate in the study.
* Angiographic exclusion criteria:

  1. Infarct artery reference vessel diameter <2.5 mm on visual assessment.
  2. Previously stented infarct artery.
  3. TIMI thrombus grade < 4.
  4. Inability to identify the infarct artery.
* Contraindications to adenosine:

  1. Second or third degree atrioventricular block
  2. Sick sinus syndrome
  3. Systolic blood pressure less than 90 mm Hg
  4. Sinus bradycardia (heart rate<40 bpm)
  5. Active bronchospastic disease with regular use of inhalers
  6. Known hypersensitivity to adenosine
* Contraindications to CMR :

  1. Cerebral aneurysm clips
  2. MRI non compatible cardiac pacemaker
  3. Implanted cardioverter-defibrillator
  4. Retained transvenous pacemaker and defibrillator leads
  5. Electronic implant or device, eg, insulin pump or other infusion pump
  6. Cochlear, otologic, or other ear implant
  7. Shunt (spinal or intraventricular)
  8. Tissue expander (eg, breast)
  9. Joint replacement (eg, hip, knee, etc)
  10. Any type of prosthesis (eg, eye, penile, etc)
  11. Known claustrophobia
  12. Body piercing jewelry
  13. Known/possible pregnancy or breast feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial Salvage Index assesed by CMR | 48 hours after the Intervention and after 3 month of the STEMI.
  Myocardial salvage index (MSI) will be determined as the difference between the area at risk and the total infarct area divided by the area at risk.

SECONDARY OUTCOMES:
ST segment resolution | after 60 minutes of the procedure
  According to pre and post- procedure ECG findings.
Corrected TIMI frame count | During the coronary angio to assess flow after the procedure.
  From the final image of the coronary angiogram.

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Interventional Cardiology, Principal Investigator — Head of Interventional Cardiology Dept., Careggi Hospital - University of Florence, Italy.; Ahmed M ElGuindy, MD, MRCP, Principal Investigator — Head of Cardiology Dept. at Aswan Heart Centre - Magdi Yacoub Heart Foundation - Aswan, Egypt.
Locations (1):
- Aswan Heart Centre - Magdi Yacoub Heart Foundation, Aswān, Aswan Governorate, Egypt